CLINICAL TRIAL: NCT07074314
Title: The Effect of Laughter Yoga on Quality of Life and Premenstrual Symptoms in Young People With Premenstrual Syndrome: A Randomized Controlled Experimental Study
Brief Title: The Effect of Laughter Yoga and Premenstrual Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırklareli University (Other)
Responsible Party: Principal Investigator, Ayca Solt Kirca, Asssociate professor, Kırklareli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KırklareliAS-15
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Premenstrual Syndrome; Quality of Life
Keywords: laughter yoga; premenstraul syndrome; qualifty of life
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Laughter Therapy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laughter yoga group (Experimental): Before starting the intervention, the researcher attended a 12-hour "Laughter Yoga Leader" course (8 hours of theory and 4 hours of Laughter Yoga Practice). Following the course, the researcher received a "Laughter Yoga" certificate. In the first stage, all participants will be asked to introduce themselves by giving their names and places of birth. Then, laughter yoga will begin with warm-up exercises and hand clapping movements. In the second stage, deep breathing exercises will be performed. After the deep breathing exercises, in the third stage, childlike games will be used to help induce laughter. In the final stage, laughter exercises will be conducted. Laughter yoga sessions will be conducted twice a week for 8 weeks, for a total of 16 sessions. Each session will be 30 minutes in duration.
  Interventions: Other: Laughter yoga
- Control group (No Intervention): Participants in this group will consist of people who do not routinely do any practice on their own to reduce stress and burnout levels. The researcher will ask the participants via phone 4 times a week for 1 month whether they have taken any action to reduce their stress and burnout symptoms. Participants who use any of the pharmacological or non-pharmacological practices to reduce stress and burnout symptoms will be excluded from the study.

INTERVENTIONS:
Other: Laughter yoga — Part 1: Deep Breathing Exercises: Raise the arms up towards the sky and take a deep breath as possible and hold the breath for 4-5 seconds. This application is repeated several times. This section takes approximately 5-10 minutes.
  Part 2: Warm-up exercises: Hands are kept parallel to each other and clapped. The tips of the fingers and palms touch each other, the acupuncture points on both hands are stimulated and the individual's energy level increases.
  Section 3: Childish Games: In this section there are childish games. These games are visualized in the mind and the participants are asked to raise their arms upwards in the shape of the letter "Y".This section takes approximately 10 minutes.
  Section 4: Laughter Exercises: Participants are given verbal guidance such as "Put your hand on your heart, feel your heartbeat, let's exhale with a smile, let's make a wish or pray" and the laughter exercise is terminated. This section takes approximately 15 minutes.
  Arms: Laughter yoga group

SUMMARY:
Premenstrual Syndrome (PMS) describes somatic, cognitive, emotional, and behavioral symptoms that occur in women during the luteal phase of the menstrual cycle and resolve with the onset of menstruation. These symptoms are common during the reproductive years. The emotional symptoms of PMS include depression, outbursts of anger, irritability, crying spells, anxiety, confusion, social withdrawal, poor concentration, insomnia, increased short sleep, and changes in sexual desire. Premenstrual symptoms negatively impact women's relationships with family, work, and friends, as well as their social activities. Furthermore, premenstrual symptoms negatively impact a woman's quality of life, making them an important issue to address early in a woman's life. Numerous treatment methods are used to reduce or eliminate PMS symptoms. Laughter yoga is one of the alternative medicine methods that has recently emerged and is used to maintain and improve health. No studies have examined the effectiveness of laughter yoga in reducing premenstrual syndrome. This study aims to determine the effects of laughter yoga on quality of life and premenstrual symptoms in young people experiencing premenstrual syndrome.

DETAILED DESCRIPTION:
Premenstrual Syndrome (PMS) describes somatic, cognitive, emotional, and behavioral symptoms that occur in women during the luteal phase of the menstrual cycle and resolve with the onset of menstruation. These symptoms are common during the reproductive years. The emotional symptoms of PMS include depression, outbursts of anger, irritability, crying spells, anxiety, confusion, social withdrawal, poor concentration, insomnia, increased short sleep, and changes in sexual desire. Physical symptoms include thirst, appetite changes, breast tenderness, bloating and weight gain, headaches, swelling in the hands or feet, aches and pains, fatigue, skin problems, and gastrointestinal symptoms, which can occur in the days before and after menstruation. While the epidemiology, etiology, and pathophysiology of PMS, first described in the literature in 1931, have not yet been fully elucidated, factors that may contribute to its development include thyroid dysfunction, hormonal changes, neurotransmitters, hypoglycemia, fluid retention, genetic and psychological factors, diet, stress, and lifestyle. Epidemiological studies indicate that PMS affects approximately one-fifth of women. Therefore, while PMS is common in adolescence and young adulthood, it stands out as a significant problem during this period. Premenstrual symptoms negatively impact women's relationships with family, work, and friends, as well as their social activities. They can lead to losses in education and employment, decreased work productivity, increased error/accident rates, alcohol/substance abuse, and criminal behavior, and negative mother-child behavior. It's also known that mental disorders and physical illnesses worsen during the premenstrual period, and psychiatric hospitalizations increase. Furthermore, premenstrual symptoms negatively impact a woman's quality of life, making them an important issue to address early in a woman's life. Numerous treatment methods are used to reduce or eliminate PMS symptoms.

The goal of treatment for PMS is to reduce or eliminate symptoms, reduce negative impacts on activities and relationships, and minimize treatment side effects. A stepwise approach should be implemented in PMS treatment, encompassing non-pharmacological treatment, pharmacological treatment, and surgical treatment. It has been reported that 60% of women with PMS symptoms seek treatment for their symptoms, but only about half as often seek medical attention.

Recommended non-pharmacological treatments include lifestyle changes, education, dietary support, herbal treatment options, acupuncture, and cognitive behavioral therapy. Lifestyle changes include regular exercise, limiting caffeine, salt, and alcohol consumption, eliminating nicotine, and increasing complex carbohydrate intake. Exercise has been shown to reduce PMS symptoms. Shifting focus is particularly important. Cognitive therapy methods and physical activity have been found to reduce PMS symptoms. Alternative medicine methods, in particular, are widely used to reduce PMS symptoms.

Laughter yoga is one of the alternative medicine methods that has recently emerged and is used to maintain and improve health. Laughter is generally considered a visual expression of happiness or a feeling of joy. It also helps clarify one's intentions in social interactions and foster emotional connection in conversations. Laughter is contagious; when a person laughs, the person next to them is often moved and begins to laugh as well. Laughter has been described as a universal phenomenon that can be observed in the body and contributes to irreplaceable social functions. During the emergence of laughter, people establish relationships between objects and attribute specific meanings to them by comparing them with others. The combination of all these factors provides relief. People laugh not only at humor, but also when solving a puzzle, escaping a dangerous situation, winning a game, experiencing disappointment, feeling hopeless, encountering an old friend, feeling embarrassed, or angry. Laughter can occur in a variety of emotional states. Laughter yoga has been found to lower cortisol levels, stabilize blood pressure, and improve quality of life scores, especially after the fourth session. Laughter yoga has been found to have a positive impact on young people's overall health, improving physical well-being and symptoms of sleep disorders, reducing anxiety and depression scores, and improving social functioning. In this context, considering the uses and benefits of laughter yoga, it is thought that it may be effective in reducing PMS symptoms. There are numerous studies in the literature on premenstrual syndrome. However, few studies have investigated the effectiveness of alternative methods for reducing symptoms. No studies have examined the effectiveness of laughter yoga in reducing premenstrual syndrome. This study aims to determine the effects of laughter yoga on quality of life and premenstrual symptoms in young people experiencing premenstrual syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research
* Fully answering survey and scale forms
* Ability to read and understand Turkish
* Being between the ages of 18 and 25 years
* Having regular menstruation (between 21 and 35 days)

Exclusion Criteria:

* Unwilling to continue working
* Having any problem that prevents communication (such as hearing, speaking, and understanding abilities),
* Having a gynecological disease (abnormal uterine bleeding, uterine fibroids, ovarian cysts, hormonal treatment, etc.)
* Having a chronic or physical illness
* Having a mental illness
* Being under psychiatric treatment (Pharmacotherapy or psychotherapy)
* Taking medication for menopausal symptoms
* Using one of the pharmacological or non-pharmacological methods to reduce premenstrual symptoms (COCs, acupressure, homeopathy, etc.)

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2025-12-25 (Actual); Primary Completion 2025-12-25 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
The Premenstrual Symptoms Coping Scale | between 2 to 4 weeks
  This scale assesses the coping with premenstrual symptoms in women aged 18-49. The scale consists of 27 items and five subscales in Turkish. Each item on this five-point Likert-type scale is scored from one to five. The total score is not used.
Premenstrual Syndrome-Specific Quality of Life Scale | between 2 to 4 weeks
  The scale consists of 22 items divided into three subscales: physical, emotional, and social. Reverse coding is used for all items, with a minimum score of 22 and a maximum score of 110.

CONTACTS AND LOCATIONS:
Overall Officials: ELIF DAGLI, Phd, Study Director — Cukurova University
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)